CLINICAL TRIAL: NCT02979665
Title: A Clinico-Pathological Study of the Structural and Functional Changes to the Retina Following Anti-VEGF Treatments for Diabetic Macular Edema
Brief Title: Changes to the Retina Following Anti-VEGF Treatments for Diabetic Macular Edema
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 105570
Record Dates: First submitted 2016-11-25; First posted 2016-12-01 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Ranibizumab Ophthalmic: DME consults requiring anti-VEGF treatment
  Interventions: Drug: Ranibizumab Ophthalmic
- Control: DME consults not requiring anti-VEGF

INTERVENTIONS:
Drug: Ranibizumab Ophthalmic — Ranibizumab (trade name Lucentis among others) is a monoclonal antibody fragment (Fab) created from the same parent mouse antibody as bevacizumab. It is an anti-angiogenic that has been approved to treat the "wet" type of age-related macular degeneration (AMD, also ARMD), a common form of age-related vision loss and diabetic macular edema (DME).
  Other Names: Lucentis
  Groups: Ranibizumab Ophthalmic

SUMMARY:
anti-VEGF therapy is an established method to control leakage and abnormal growth of retinal blood vessels. Questions on the long-term effect on the retina, intraocular pressure and on the overall retinal perfusion from these treatments remain to be answered. The purpose of the study was to evaluate changes in the retina following anti-VEGF treatment over time, using structural and functional diagnostic tests.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) causes changes in the capillaries that nourish the retina. Two treatments clinically used for DR are laser photocoagulation to reduce the angiogenic drive by knocking off metabolically active retina and anti-VEGF drugs for diabetic macular edema (DME). DME affects approximately 2.5% of the nearly 2.4 million Canadians with diabetes, or approximately 60,000 Canadians, making it a major cause of adult-onset vision loss. DME occurs when blood vessels in the retina of diabetic patients become leaky resulting in unwanted fluid accumulation in the center of vision known as the macula. If not treated, this can lead to blindness. Originally used in the treatment of age-related macular degeneration (AMD), anti-VEGF drugs are increasingly used to control leakage and abnormal growth of retinal blood vessels. Numerous questions have emerged following the usage of anti-VEGF medications in the eye such as their long-term effects of these drugs on intraocular pressure and on the overall retinal perfusion. By recruiting DR patients requiring anti-VEGF treatment for DME, this study will answer whether long-term usage of anti-VEGF will result in structural and functional changes to the retina.

ELIGIBILITY:
Inclusion Criteria:

* DME patients
* Require anti-VEGF injections in at least one eye

Exclusion Criteria:

* Advanced lens opacity or cataract that could affect diagnostic testing
* Prior retinal treatment (PRP, focal laser or surgery within 6 months of participation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DR consults referred to the Ivey Eye Institute and requiring anti-VEGF injections in at least one eye due to DME will be recruited into the study.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Effects of anti-VEGF drugs on intraocular pressure (mmHg) | 2 year

SECONDARY OUTCOMES:
Effects of anti-VEGF drugs on macular thickness (um) | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Hutnik, MD, PhD, Principal Investigator — St. Joseph's Health Care London

REFERENCES:
- [Background] Simo R, Hernandez C. Intravitreous anti-VEGF for diabetic retinopathy: hopes and fears for a new therapeutic strategy. Diabetologia. 2008 Sep;51(9):1574-80. doi: 10.1007/s00125-008-0989-9. Epub 2008 Apr 11. PMID 18404258
- [Background] Osaadon P, Fagan XJ, Lifshitz T, Levy J. A review of anti-VEGF agents for proliferative diabetic retinopathy. Eye (Lond). 2014 May;28(5):510-20. doi: 10.1038/eye.2014.13. Epub 2014 Feb 14. PMID 24525867
- [Background] Singh RS, Kim JE. Ocular hypertension following intravitreal anti-vascular endothelial growth factor agents. Drugs Aging. 2012 Dec;29(12):949-56. doi: 10.1007/s40266-012-0031-2. PMID 23179897
- [Background] Mathalone N, Arodi-Golan A, Sar S, Wolfson Y, Shalem M, Lavi I, Geyer O. Sustained elevation of intraocular pressure after intravitreal injections of bevacizumab in eyes with neovascular age-related macular degeneration. Graefes Arch Clin Exp Ophthalmol. 2012 Oct;250(10):1435-40. doi: 10.1007/s00417-012-1981-0. Epub 2012 Mar 21. PMID 22434210
- [Background] Neubauer AS, Kook D, Haritoglou C, Priglinger SG, Kampik A, Ulbig MW, Ceklic L. Bevacizumab and retinal ischemia. Ophthalmology. 2007 Nov;114(11):2096. doi: 10.1016/j.ophtha.2007.05.057. No abstract available. PMID 17980746
- See also: Canadian Diabetes Association. Eye Damage (Diabetic Retinopathy). — http://www.diabetes.ca/diabetes-and-you/complications/eye-damage-diabetic-retinopathy